CLINICAL TRIAL: NCT06340737
Title: Phase Ib Clinical Trial of Autologous CD22 Chimeric Antigen Receptor (CAR) T Cells in Adults With Recurrent or Refractory B Cell Lymphomas
Brief Title: AutologousCD22 Chimeric Antigen Receptor (CAR)T Cells in w/Recurrent/Refractory B Cell Lymphomas
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: The Leukemia and Lymphoma Society (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-73394; NCI-2024-03048 (Registry Identifier: NCI- Clinical Trial Reporting Program)
Record Dates: First submitted 2024-03-08; First posted 2024-04-01 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Follicular Lymphoma; Mantle Cell Lymphoma; Hairy Cell Leukemia; Lymphoplasmacytic Lymphoma; Burkitt Lymphoma; Marginal Zone Lymphoma; Waldenstrom Macroglobulinemia; Large B-cell Lymphoma
Keywords: lymphoma; leukemia; lymphodepleting chemotherapy; relapsed; refractory; systemic therapy
MeSH Terms: conditions — Lymphoma, Follicular; Lymphoma, Mantle-Cell; Leukemia, Hairy Cell; Lymphoma, B-Cell, Marginal Zone; Burkitt Lymphoma; Waldenstrom Macroglobulinemia; Lymphoma; Leukemia; Recurrence

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1: Follicular lymphoma (FL) (Experimental): 18-34 participants with FL will be administered the RP2D of CD22CART
  Interventions: Drug: CD22CART Infusion
- Cohort 2: Mantle cell lymphoma (MCL) (Experimental): 12-32 participants with MCL will be administered the RP2D of CD22CART.
  Interventions: Drug: CD22CART Infusion
- Cohort 3: Other lymphomas (Experimental): Up to 30 participants with no more than 10 of any one type, including: Hairy cell leukemia, Lymphoplasmacytic lymphoma (Waldenstrom macroglobulinemia), Burkitt lymphoma, and Marginal zone lymphoma.
  Interventions: Drug: CD22CART Infusion
- Cohort 4: Relapsed/refractory large B cell lymphoma (LBCL) (Experimental): 14 - 19 participants will be administered the RP2D of CD22 CART
  Interventions: Drug: CD22CART Infusion

INTERVENTIONS:
Drug: CD22CART Infusion — Dosing and Administration Participants will be hospitalized to receive treatment with CD22CART, if not previously hospitalized, and will remain hospitalized for approximately 5 to 7 (±2) days. Patients may be discharged once all AEs have resolved to Grade 1 or better, or at the discretion of the treating physician. Participants may be discharged with non critical and clinically stable or slowly improving toxicities (e.g., renal insufficiency, cytopenias) even if > Grade 1, if deemed appropriate by the investigator.

SUMMARY:
This is a non-randomized clinical trial to evaluate the safety and efficacy of CD22CART administered after lymphodepleting chemotherapy in adults with relapsed / refractory B Cell Lymphomas. All evaluable participants will be followed for overall survival (OS), progression free survival (PFS), and duration of response (DOR). An evaluable participant is one who completes leukapheresis, lymphodepleting chemotherapy and CART infusion.

ELIGIBILITY:
Inclusion Criteria:

* Disease: Must have histologically confirmed disease as defined by WHO 2016[117] of one of the following:

Follicular Lymphoma, grade 1-3a

1. Relapsed or refractory disease after at least 2 lines of systemic therapy. Prior therapy must have included an anti-CD20 monoclonal antibody combined with systemic therapy (single-agent anti- CD20 antibody does not count as line of therapy for eligibility nor does local radiation). Anti-CD20 antibody is not required for participants with CD20 negative disease. A systemic therapy includes, but is not limited to: Bendamustine, CHOP, CVP, CART therapy, lenalidomide, or platinum-based chemotherapy.
2. Relapsed or progressive disease within 24 months of initiation of the initial course of chemotherapy (also known as progression of disease within 24 months POD24). Initial treatment must have included an anti-CD20 monoclonal antibody (unless CD20 negative) plus either Bendamustine, CHOP or CVP (R-Chemo). Must have completed 3 or more cycles of R-Chemo. Progression is measured from the initial day of treatment of the first cycle of R-Chemo. In the case of those who received anti-CD20 monoclonal antibody monotherapy previously and then received R-Chemo are also eligible if they are POD24, and progression is measured from the initial day of treatment of the first cycle of R-Chemo and not from the initial day of anti-CD20 monoclonal antibody monotherapy.

Mantle Cell Lymphoma 1. Relapsed or refractory disease after at least 2 lines of systemic therapy. Prior therapy must have included an anti-CD20 monoclonal antibody combined with systemic therapy. Anti-CD20 antibody is not required for participants with CD20negative disease.

2. Participants who have received an anti-CD20 monoclonal antibody in combination with chemotherapy AND a Bruton's Tyrosine Kinase inhibitor as a single line of therapy are also eligible.

Hairy cell leukemia (HCL)

1. Diagnosis of HCL and require treatment as defined by having HCL-related anemia (hemoglobin <11 g/dL), thrombocytopenia (platelets<100 x 10^9 /L), or neutropenia (absolute neutrophil count below 1.5 x 10^9/L); symptomatic splenomegaly or adenopathy; or other constitutional symptoms directly related to HCL;
2. Must have progressed or been refractory to 2 lines of therapy including a purine nucleoside analog.

Lymphoplasmacytic lymphoma (Waldenstrom macroglobulinemia (WM)) - participants must meet all eligibility criteria listed

1. Must have confirmed diagnosis of WM based on Second International Workshop on WM 2. Relapsed or refractory disease after 2 or more lines of therapy

1. Prior therapies must include a i. BTKi ii. either chemotherapy and/or proteasome inhibitor 3. Requires treatment based on the recommendations from the Second International Workshop on WM 4. Requires the presence of serum IgM that is at least 2 times the upper limit of normal 5. Patients cannot require plasmapheresis for symptomatic hyperviscosity. 6. Patients cannot have symptomatic central nervous system involvement (Bing-Neel syndrome) that would prevent the assessment of neurotoxicity 7. Patients cannot have transformed to large B cell lymphoma Burkitt lymphoma (BL)

1. Relapsed or refractory to front line chemoimmunotherapy; Participants with high-grade B-cell lymphoma with MYC and BCL2 and/orBCL6 rearrangements will be excluded.

Marginal zone lymphoma (MZL)

1. Must have received 2 prior lines of therapy including rituximab in combination with chemotherapy or a BTKi

Histologically confirmed Large B-cell lymphoma (LBCL) by WHO 2008 including:

i. DLBCL not otherwise specified; DLBCL associated with chronic inflammation; Epstein Barr virus (EBV)+ DLBCL of the elderly; OR ii. primary mediastinal (thymic) large B cell lymphoma; OR iii. transformation of follicular lymphoma, marginal zone lymphoma or chronic lymphocytic leukemia/small lymphocytic lymphoma to DLBCL; OR iv. Follicular Lymphoma Grade 3B

• Subjects with DLBCL, Follicular Lymphoma Grade 3B -or-

Subjects with transformed FL and MZL who HAVE NOT received chemotherapy prior to transformation:

1) Must have received an anthracycline regimen and an anti CD20 monoclonal antibody (unless documented CD20-negative) and be refractory or relapsed after second line of LBCL treatment. Subjects with a partial response to second line therapy must be ineligible for autologous transplant.

* Subjects with transformed FL and MZL who HAVE received anthracycline-containing chemotherapy prior to transformation must have progressed, had SD or recurred with transformed disease after initial treatment for LBCL:

  1. Must have progressed, had SD, or recurred with transformed disease after initial treatment for LBCL

     Note: T cell/histiocyte rich large B cell lymphoma is not eligible

     The following criteria apply to all participants unless otherwise noted:

  2. Measurable Disease:
  1. a. Participants with Follicular Lymphoma, Mantle Cell Lymphoma, Burkitt Lymphoma and Marginal Zone Lymphoma must have measurable disease according to the revised IWG Response Criteria for Malignant Lymphoma. Lesions that have been previously irradiated will be considered measurable only if progression has been documented following completion of radiation therapy.

     b. If participants with Follicular Lymphoma, Mantle Cell Lymphoma, Burkitt Lymphoma, Marginal Zone Lymphoma, and Large B cell Lymphoma that do not have measurable disease according to the revised IWG Response Criteria for Malignant Lymphoma, but have disease that is greater than 2% of events by flow cytometry in the peripheral blood or bone marrow will be eligible
  2. c. Participants with Hairy Cell Lymphoma must have presence of leukemic cells in the bone marrow or blood stream.
  3. d. Participants with Lymphoplasmacytic lymphoma must have the presence of serum IgM that is at least 2 times the upper limit of normal.

  3. CD22 expression, at any level: Participants must have archival tissue available for analysis of CD22 expression or must be willing to undergo biopsy of easily accessible disease.

  4. Participants who have progressed or relapsed after prior autologous OR allogeneic SCT must be at least 100 days post-transplant, have no evidence of GVHD, and have been without immunosuppressive drugs at least 30 days.

  5. Meet required prior therapy washout windows prior to leukapheresis (see inclusion criteria for leukapheresis for details).

  6. Participants with prior CAR therapy must be at least 30 days post CAR infusion and have < 5% CD3+ cells express the previous CAR prior to apheresis, if a validated assay is available.

  7. Toxicities from prior therapy stable or resolved (except for clinically non-significant toxicity and cytopenias covered in footnote).

  8. Age ≥ 18 years of age. 9. Adequate performance status (ECOG 0, 1, or 2; or Karnofsky > 60%) 10. Adequate organ and marrow function as defined by:

  - ANC ≥ 750/uL
  * Platelet count ≥ 50,000/uL
  * ALC ≥ 150/uL
  * Adequate renal, hepatic, pulmonary and cardiac function defined as: Creatinine < 2 mg/dL OR Creatinine clearance (as estimated by Cockcroft Gault Equation) ≥ 45 mL/min, Serum ALT or AST ≤ 10 x ULN (except in participants with liver involvement by lymphoma), Total bilirubin ≤ 1.5 mg/dl, except in participants with Gilbert's syndrome, Cardiac left ventricular ejection fraction ≥ 45%, no evidence of clinically significant pericardial effusion as determined by an Echocardiogram.
  * No clinically significant pleural effusion or ascites
  * Baseline oxygen saturation > 92% on room air ANC Platelet ALC Cr CreatCl AST/ALT Bilirubin LVEF O2 Sat
  * 11. Participants with CNS involvement or a history of CNS involvement are eligible only in the absence of neurologic symptoms that may mask or interfere with neurological assessment of toxicity 12. Females of childbearing potential must have negative pregnancy test. 13. Females of child-bearing potential and males of child-fathering potential must be willing to practice birth control from time of enrollment and for 4 months post preparative lymphodepletion regimen or as long as CAR cells are detectable.

    14. Must be able to provide informed consent (LAR is permitted if participant able to provide verbal assent).

A participant will not be excluded because of pancytopenia ≥ Grade 3 if it is felt by the investigator to be due to underlying disease.

Exclusion Criteria:

* Presence rapidly progressive disease that in the estimation of the investigator and sponsor would compromise ability to complete study therapy.

  2. History or current other malignancies, apart from non-melanoma skin cancer, low-grade untreated prostate cancer under observation, or carcinoma in situ, unless disease free for at least 3 years, or in remission 1-2 years and Principal Investigator assesses other malignancy as unlikely to return within 1 year or interfere with CAR T cell safety

  3. Presence of active fungal, bacterial, viral or other infection requiring intravenous antimicrobials. Simple UTI or uncomplicated bacterial pharyngitis is permitted if responding to active treatment.

  4. Ongoing HIV, HBV, or HCV infection. History of HBV or HCV is permitted if viral load is undetectable by qPCR and/or nucleic acid testing.

  5. Active cerebrovascular ischemic/hemorrhage, dementia, cerebellar disease, or autoimmune disease with CNS involvement that in investigator's judgement impair ability to evaluate neurotoxicity.

  6. History of MI, cardiac angioplasty or stenting, unstable angina or other clinically significant cardiac disease within 12 months of enrollment.

  7. Severe, immediate hypersensitivity reaction attributed to compounds of similar chemical or biologic composition to any agents used in study.

  8. Is pregnant or breastfeeding.

  9. Active primary immunodeficiency or history of autoimmune disease (e.g. Crohn's disease, rheumatoid arthritis, systemic lupus) requiring systemic immunosuppression/systemic disease modifying agents within the last 2 years.

  10. May NOT, in investigator's judgment, have any medical condition likely to interfere with assessment of safety or efficacy, or be likely to complete all protocol-required visits and procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Estimated)
Dates: Start 2024-03-29 (Actual); Primary Completion 2031-04 (Estimated); Study Completion 2031-04 (Estimated)

PRIMARY OUTCOMES:
Determine the manufacturing feasibility of CD22 CART by assessing the target dose level and release specifications in each disease cohort. | 6 years
  Rate of successful manufacture of CD22CART cells at the target dose level that meet required release specifications in Cohort 1, Cohort 2, and Cohort 3.
Maximum tolerated dose (MTD)/recommended phase 2 dose (RP2D) | 6 years
  Establish the maximum tolerated dose (MTD)/recommended phase 2 dose (RP2D) of CD22CART cells in 3 cohorts of adults with relapsed/refractory B Cell lymphoma.
Determine the overall response rate (ORR) in adults with follicular lymphoma (FL) and mantle cell lymphoma (MCL) | 3 months CD22 CART infusion
  Assess the ORR at 3 months post CD22 CART infusion as defined by the disease specific response criteria for Cohort 1 (FL) and Cohort 2 (MCL)

SECONDARY OUTCOMES:
Evaluate Progression Free Survival (PFS) | 6 years
  Evaluate Progression Free Survival (PFS) in adults with relapsed/refractory B cell lymphoma after receiving CD22CART. PFS defined as the interval from CD22CART infusion to time of disease progression or death from any cause
Evaluate Overall Survival (OS) | 6 years
  Evaluate Overall Survival (OS) in adults with relapsed/refractory B cell lymphoma after receiving CD22CART. OS defined as the interval from CD22CART infusion to the time of death from any cause.
Evaluate Duration of Response (DOR) | 6 years
  Evaluate Duration of Response (DOR) in adults with relapsed/refractory B cell lymphoma after receiving CD22CART. DOR defined as the interval from achieving an objective response to the time of disease progression.
Assess the response rate in adults with relapsed/refractory Hairy cell leukemia (HCL), Lymphoplasmacytic lymphoma (Waldenstrom macroglobulemia) (WM), Burkitt lymphoma (BL), and Marginal Zone lymphoma (MZL). | 3 months post CD22
  Describe the response rates assessed at 3 months post CD22 CART infusion for Cohort 3 (HCL, WM, BL, and MZL).

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Frank, MD, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Palo Alto, California, United States